CLINICAL TRIAL: NCT05070078
Title: The Single Assessment Numeric Evaluation (SANE): Is a Reliable Metric to Measure Clinically Significant Improvements After Lumbar Discectomy
Brief Title: The Single Assessment Numeric Evaluation (SANE) for Lumbar Discectomy
Status: Recruiting | Type: Observational
Sponsor: Windsor-Essex Compassionate Care Community (Other)
Responsible Party: Principal Investigator, Mohamed Soliman, Neurosurgeon, Principal Investigator, Windsor-Essex Compassionate Care Community
Other Study IDs: 21-409
Record Dates: First submitted 2021-09-05; First posted 2021-10-06 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Lumbar Discectomy
Keywords: Lumbar Discectomy; Single Assessment Numeric Evaluation; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the last several decades, many Patient Reported Outcomes Measures (PROMs) have been developed to provide assessment of patient health across multiple domains, as they relate to various spine conditions. However, many of the available PROM surveys have many questions and require substantial time to complete and/or assess one focal domain of health requiring multiple tools to achieve an overall assessment of well-being. Thus, concerns have arisen regarding patient survey fatigue and data integrity.

The Single Assessment Numeric Evaluation (SANE) is a single-question outcome measure that asks patients to rate their function, as it pertains to the area being treated, on a scale of 0 to 100. The SANE score has excellent acceptance in some orthopedic surgery research, where it has been shown responsiveness similar to more comprehensive legacy measures. The SANE thus eliminates survey fatigue and has been validated across a spectrum of orthopedic subspecialties. To our knowledge, however, the SANE has never been studied in a patient population undergoing any type of spinal surgery. Thus, we set out to compare the SANE score in patients undergoing lumbar discectomy to currently utilized PROM scores, including the Oswestry Disability Index (ODI), Zurich Claudication Scale (ZCS), and short form-36 (SF-36).

DETAILED DESCRIPTION:
Background/Rational: In the last several decades, many Patient Reported Outcomes Measures (PROMs) have been developed to provide assessment of patient health across multiple domains, as they relate to various spine conditions. When considered in concert, these instruments quantify and stratify an individual's health state before and after surgery and can be utilized to perform research as well as inform clinical practice. However, many of the available PROM surveys have many questions and require substantial time to complete and/or assess one focal domain of health requiring multiple tools to achieve an overall assessment of well-being. Thus, concerns have arisen regarding patient survey fatigue and data integrity. Ideally, a PROM would provide sufficient information to define health status longitudinally, while requiring the least amount of time and effort to complete. The current approach to PROMs in spine surgery research has been mostly to require an assessment of pain, disease specific disability and general health, requiring answers for up to of 40 unique questions, despite efforts to shorten the questionnaires in other neurosurgery and orthopedics disciplines.

The Single Assessment Numeric Evaluation (SANE) score is one such example of a limited question survey that aims to assess multiple domains. The SANE is a single-question outcome measure that asks patients to rate their function, as it pertains to the area being treated, on a scale of 0 to 100. The SANE score has excellent acceptance in some orthopedic surgery research, where it has been shown responsiveness similar to more comprehensive legacy measures. The SANE thus eliminates survey fatigue and has been validated across a spectrum of orthopedic subspecialties. To our knowledge, however, the SANE has never been studied in a patient population undergoing any type of spinal surgery. Thus, we set out to compare the SANE score in patients undergoing lumbar discectomy to currently utilized PROM scores, including the Oswestry Disability Index (ODI), Zurich Claudication Scale (ZCS), and short form-36 (SF-36).

Design: Survey research design, prospective outcomes measure validation study.

Objectives: We hypothesized that the SANE score would correlate strongly and demonstrate similar magnitudes of longitudinal responsiveness with the more lengthy and burdensome legacy PROMs used in spine surgery research today.

Primary Objective: To correlate and confirm that SANE score to the more lengthy and burdensome legacy PROMs used in spine surgery research today.

Secondary Objective: There are multiple secondary aims of this study as shown below.

1. Evaluate patients' satisfaction after surgery.
2. Assess efficacy of treatment over time.
3. Evaluate patients' sense of functional improvement after lumbar disc procedures.

Information gained from this study will greatly enhance our ability to know whether SANE correlates with PROMS. Although the results of the trial will not directly benefit all the individuals participating, information gathered from this study can help future patients by reducing the burden of completing lengthy surveys and minimizing survey fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age undergoing a lumbar discectomy.

Exclusion Criteria:

* Previous history of lumbar surgery.
* Pediatric age group.
* Patients with a postoperative follow-up time of less than 1 year.
* Unstable patients in need of fixation.
* Patients with cauda equina syndrome.
* Non-compliant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lumbar discectomy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2028-12-10 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Correlation of SANE score | November 2022
  To correlate and confirm that SANE score to the more lengthy and burdensome legacy PROMs used in spine surgery research today. Spearman's correlation and linear regression will be performed for each time point, and for the change from preoperative to final follow up to validate the SANE as compared to the other PROMs.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Soliman, Principal Investigator — Cairo University
Locations (1):
- Windsor Regional Hospital - Ouellette, Windsor, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shelbourne KD, Barnes AF, Gray T. Correlation of a single assessment numeric evaluation (SANE) rating with modified Cincinnati knee rating system and IKDC subjective total scores for patients after ACL reconstruction or knee arthroscopy. Am J Sports Med. 2012 Nov;40(11):2487-91. doi: 10.1177/0363546512458576. Epub 2012 Sep 12. PMID 22972851
- [Background] Stokes OM, Cole AA, Breakwell LM, Lloyd AJ, Leonard CM, Grevitt M. Do we have the right PROMs for measuring outcomes in lumbar spinal surgery? Eur Spine J. 2017 Mar;26(3):816-824. doi: 10.1007/s00586-016-4938-x. Epub 2017 Jan 9. PMID 28070683
- [Background] Weinstein JN, Tosteson TD, Lurie JD, Tosteson AN, Hanscom B, Skinner JS, Abdu WA, Hilibrand AS, Boden SD, Deyo RA. Surgical vs nonoperative treatment for lumbar disk herniation: the Spine Patient Outcomes Research Trial (SPORT): a randomized trial. JAMA. 2006 Nov 22;296(20):2441-50. doi: 10.1001/jama.296.20.2441. PMID 17119140
- [Result] Torchia MT, Austin DC, Werth PM, Lucas AP, Moschetti WE, Jevsevar DS. A SANE Approach to Outcome Collection? Comparing the Performance of Single- Versus Multiple-Question Patient-Reported Outcome Measures After Total Hip Arthroplasty. J Arthroplasty. 2020 Jun;35(6S):S207-S213. doi: 10.1016/j.arth.2020.01.015. Epub 2020 Jan 16. PMID 32008770